CLINICAL TRIAL: NCT06666751
Title: Post-operative Anterior Segment OCT Evaluation of Trabecular Microstent Positioning and the Impact on Intraocular Pressure
Brief Title: Anterior Segment Optical Coherence Tomography Microstent Positioning
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Rachel Simpson, Assistant Professor (Clinical), University of Utah
Other Study IDs: 163214
Record Dates: First submitted 2024-10-21; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Glaucoma; Stent Migration; Stent Dislodgement; Intraocular Pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hydrus microstent: Participants in this group underwent Hydrus microstent placement at the Moran Eye Center.
  Interventions: Procedure: Cataract plus Microstent surgery
- iStent Inject: Participants in this group underwent iStent Inject placement at the Moran Eye Center.
  Interventions: Procedure: Cataract plus Microstent surgery

INTERVENTIONS:
Procedure: Cataract plus Microstent surgery — Both the Hydrus microstent and iStent Inject W are used in combination with cataract surgery, in order to help lower intraocular pressure for patients with open-angle glaucoma. The microstent is a small flexible device that is inserted into the eye during cataract surgery in order to improve the outflow of fluid from the eye.

SUMMARY:
The goal of this observational study is to learn about the long-term results of glaucoma stent surgery in men and women 18 or older who have had cataract and microstent surgery in the past 2 years at the Moran Eye Center. The main questions the study aims to answer are:

1. How often are microstents mispositioned?
2. What effect does microstent positioning have on intraocular pressure after surgery?

Participants will have a one-time clinic visit for an eye exam and Optical Coherence Tomography (OCT) .

From the eye exam and OCT, Researchers will assess and categorize the position of the microstents and assess the Schlemm's canal dilation.

Researchers will review the participants' medical records to acquire 2-year data for the following:

1. Surgeon type and level of experience (resident, fellow, attending ophthalmologist)
2. Proportions of proper gonioscopic placement intraoperatively for each surgeon group
3. Effectiveness of surgery, based on change in intraocular pressure (IOP) from baseline medicated IOP, number of IOP-lowering medications the patient was able to discontinue, and rate of need for additional glaucoma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any adult glaucoma patient (age 18+) who underwent Hydrus microstent or iStent Inject placement at the Moran Eye Center.

Exclusion Criteria:

* Any patient who subsequently had to have their stent removed for any reason, any patient with a history of trauma to the anterior segment or reconstruction altering typical anatomy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comes from the Moran Eye Center, which is part of an academic teaching hospital and includes multiple community clinic locations.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Difference in percentage of mispositioned stents between Hydrus microstent and iStent groups | Two years post stent placement
  Positioning of each participant's stent(s) will be evaluated by anterior segment OCT at the one-time clinical study visit.
  iStent Inject W mispositions are defined as: microstent protrusion (entire conical head not within canal), stent completely buried in the trabeculae, or not seen (i.e. 0 or only 1 stent). If the iStent position is located but the examiner is unsure if it is positioned correctly, it will be counted as misposition. If the iStent is not seen, an in office gonioscopy will be performed to confirm results. Visualization of three stents is not considered a misposition.
  Hydrus mispositions are defined as: distal tip not in canal, at least 1 window not in canal, or trabecular microstent not within transition zone.
  The between group difference of mispositioned stents will be calculated in percentage.

SECONDARY OUTCOMES:
Dilation of Schlemm's canal | Two years post stent placement
  The Schlemm's canal is a circular lymphatic-like vessel in the eye that maintains fluid homeostasis by draining aqueous humor from the eye into the systemic circulation. If the canal is blocked, the pressure in the eye can increase, resulting in glaucoma. Dilation will be visualized on OCT and graded on a numerical scale 1-3 (1=dilated, 2=some dilation, 3=no dilation) at the one-time study visit.
Change in IOP from baseline | Two years post stent placement
  IOP is measured in millimeters of mercury (mmHg). A retrospective chart review will be conducted to acquire 2-year data to determine the change in each participant's IOP from baseline. The between group difference of change in IOP will be calculated in percentage.
Reduction in number of IOP lowering medications | Two years post stent placement
  A retrospective chart review will be conducted to determine how many IOP lowering medications each patient is using at 2 years post-stent placement compared to the number of IOP lowering medications they were using prior to stent placement. The between group difference of reduction in number of medications will be calculated in percentage.
Percentage of patients needing additional glaucoma surgery | Two years post stent placement
  A retrospective chart review will be conducted to determine the percentage of patients who had additional glaucoma surgery by the two-year post stent placement timepoint. The between group difference in number of patients needing additional glaucoma surgery will be calculated in percentage.
Sub-analysis of primary outcome by surgeon type | Two years post stent placement
  There will be a sub-analysis of the percentage of mispositions (primary endpoint) by level of surgeon experience. A retrospective chart review of the intraoperative note will determine if the primary surgeon was a resident or non-resident (attending or fellow).
Proportion of stent cases with proper placement via anterior segment OCT versus proportion of cases with proper placement via intraoperative gonioscopy | Two years post stent placement
  The intraoperative notes at the time of stent placement will include confirmation of proper stent placement via gonioscopy. At the time of the study visit, stent placement will be assessed via anterior segment OCT. The number of correctly positioned stent placements will be reported in percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Simpson, MD, Principal Investigator — Moran Eye Center
Locations (1):
- Moran Eye Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No